CLINICAL TRIAL: NCT05806775
Title: Feasibility of Low-load Resistance Training With Blood Flow Restriction in People With Advanced Disability Due to Parkinson's Disease
Brief Title: Low-load Resistance Training With Blood Flow Restriction in People With Parkinson's Disease
Acronym: BFR-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Davis Phinney Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2333
Record Dates: First submitted 2023-03-24; First posted 2023-04-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Blood Flow Restriction; Low-load resistance training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-load resistance training with blood flow restriction (Experimental): Exercises will target bilateral 1) knee extensor, 2) ankle plantarflexor, and 3) elbow extensor muscles. Exercises will be dosed based on 1RM and individualized for each participant from a standardized exercise set. Progression will be based on 1) body position (supine, seated, standing), and 2) degree of resistance. Dosing will be re-assessed every 2 weeks and progressed as tolerated. Resistance will be provided by the Shuttle Mini-Press (Shuttle Systems), a portable resistance trainer that allows for precise dosing but is also adaptable to people with mobility limitations.
  Interventions: Behavioral: Low-load resistance training with blood flow restriction

INTERVENTIONS:
Behavioral: Low-load resistance training with blood flow restriction — A licensed physical therapist, will deliver intervention to all participants (2x/wk, 8 wks) using an FDA-cleared BFR system, the Delfi PTSII (Delfi Medical Innovations). The pressure cuff will be placed at the most proximal portion of the limb and dosed following standard BFR guidelines: 1 set of 30 reps, then 3 sets of 15 reps at 20-30% 1RM with a minimum of 60% and a maximum of 80% limb occlusion pressure. At 60-80% limb occlusion pressure there is diminished venous outflow to induce the necessary metabolic effect while still allowing arterial flow for safety. Individual limb occlusion pressures will be determined at the beginning of each session automatically by the Delfi PTSII device.

SUMMARY:
The study's objective is to determine the feasibility of low-load resistance training with blood flow restriction in people who have advanced Parkinson's disease and impaired mobility using a mixed-methods convergent parallel design in a single cohort. The study's long-term goal is to develop clinically feasible exercise interventions that are effective at improving mobility, participation, and quality of life for people with advanced Parkinson's disease.

DETAILED DESCRIPTION:
This study will use a mixed-methods convergent parallel design to determine the feasibility of low-load BFR training in 20 people with advanced PD symptoms and impaired mobility (Hoehn and Yahr Stage [H&Y] 3-4). All participants will receive low intensity resistance training (20-30% of 1RM) with BFR targeting knee extensor, ankle plantarflexor, and elbow extensor muscles 2x/week for 8 weeks. Intervention will be delivered by a physical therapist with specialized training in BFR. Pre-defined feasibility criteria will be assessed in the primary aim. Outcomes assessed before and immediately after the 8-week intervention will include quantitative muscle strength and mobility assessments, and quantitative and qualitative data on health-related QOL.

Aim 1: Determine low-load BFR training feasibility based on the following quantitative and qualitative criteria: 1) enrolling 20 participants, 2) retaining ≥80% participants, 3) obtaining ≥80% intervention adherence, 4) having no serious intervention-related adverse events, and 5) quantitatively and qualitatively measured acceptability.

Aim 2: Determine changes in 1) knee extensor, ankle plantarflexor, and elbow extensor muscle strength using fixed myometry and 2) instrumented functional mobility (30-second Sit-to-Stand, Timed up and Go, self-selected walking speed, and Berg Balance Scale) using a system of inertial measurement unit wearable sensors.

Exploratory Aim: Understand health-related QOL changes using the Parkinson's Disease Questionnaire-39 (PDQ-39) and semi-structured interviews to elucidate how components of the intervention translate into QOL changes through a mixed-method analysis of PDQ-39 constructs of mobility, activities of daily living, emotional well-being, social stigma, social support, cognition, communications, and bodily discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-89 with neurologist-confirmed diagnosis of PD
* H&Y Stage 2 (bilateral involvement without postural instability) up to H&Y Stage 4 (severe disease)
* Able to provide informed consent

Exclusion Criteria:

* H&Y Stage 1 (unilateral involvement only) or less
* H&Y Stage 5 (wheelchair or bed bound)
* Unable to provide consent or diagnosis of dementia
* History of deep venous thrombosis/pulmonary embolism, peripheral vascular disease, thrombophilia or other clotting disorders; report of easy bruising
* Any comorbid conditions or pain that substantially affects ability to safely complete rehabilitation (e.g. neurologic, vascular, cardiac problems, orthopedic, or ongoing medical treatments) as determined by a neurologist or physical therapist
* Currently undergoing supervised resistance training with a physical therapist or other exercise professional
* Using Blood Flow Restriction currently or in the previous 3 months prior to enrollment
* Cannot tolerate BFR pressure cuff inflated to 60% of total limb occlusion pressure during baseline assessment
* PD-related medication change in the month prior to enrollment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Change in Knee Extension | Measured at Baseline (Week 0) and Post Test (Week 9)
  Knee extension muscle strength measured using fixed myometry (QMA Muscle Testing System)
Change in Ankle Plantarflexion | Measured at Baseline (Week 0) and Post Test (Week 9)
  Ankle plantarflexion muscle strength measured using fixed myometry (QMA Muscle Testing System)
Change in Elbow Extension | Measured at Baseline (Week 0) and Post Test (Week 9)
  Elbow extension muscle strength measured using fixed myometry (QMA Muscle Testing System)

SECONDARY OUTCOMES:
Change in 30-second Sit-to-stand Completions | Measured at Baseline (Week 0) and Post Test (Week 9)
  Functional mobility test measuring the number of sit to stand cycles a participant can complete in 30 seconds
Change in Timed Up and Go Time | Measured at Baseline (Week 0) and Post Test (Week 9)
  Functional mobility test measuring the time required to stand from sitting, walk 10 feet, turn and return to seated position at starting point
Change in Self-Selected Walking Speed | Measured at Baseline (Week 0) and Post Test (Week 9)
  Gait speed measured over a 10-meter walking course, measured in seconds
Change in Berg Balance Scale | Measured at Baseline (Week 0) and Post Test (Week 9)
  Functional mobility test measuring the participant's ability to balance in different postures. Scores on the Berg Balance Scale range from 0 to 56 points, with 0-20 points indicating wheelchair bound, 21-40 indicating walking with assistance, and 41-56 indicating walking independently.

OTHER OUTCOMES:
Change in Step Count | Measured at Baseline (Week 0) and Post Test (Week 9)
  10-day average step count as measured by a wearable activity monitor
Change in Parkinson's Disease Questionnaire-39 Score | Measured at Baseline (Week 0) and Post Test (Week 9)
  39 item questionnaire measuring quality of life in people with Parkinson's disease. Scores range from 0 to 100 with lower scores indicating higher quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No